CLINICAL TRIAL: NCT05920941
Title: Mass Balance Study of [14C]JAB-21822 in China Healthy Subjects
Brief Title: Mass Balance Study of [14C]JAB-21822
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JAB-21822-1008
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Mass Balance Study in Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]JAB-21822 (Experimental): Single oral dose of 800mg 14C]JAB-2182 suspension
  Interventions: Drug: [14C]JAB-21822

INTERVENTIONS:
Drug: [14C]JAB-21822 — Single oral administration of Carbon-14 labeled JAB-21822 800 mg/100 μCi on empty stomach

SUMMARY:
Mass Balance Study of [14C]JAB-21822 in China Healthy Subjects

DETAILED DESCRIPTION:
A phase I study to quantify the total mass balance in healthy subjects after a single dose of [14C]JAB-21822

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 45 years (inclusive).
2. Subjects weighing ≥ 50 kg and Body Mass Index of 19.0 to 26.0 kg/m2.
3. Subjects who have voluntarily participated in the study and signed the informed consent form with good compliance.

Exclusion Criteria:

1. With abnormal and clinically significant comprehensive physical examinations, vital signs, or laboratory examinations.
2. Has a positive test for HBV, HCV, HIV, or syphilis.
3. Known medical history judged by the investigator as not suitable for the study.
4. Known history of drug or food allergy.
5. Has drug or alcohol abuse history or positive drug or alcohol abuse test results.
6. Heavy smokers or caffeine addicts.
7. Has diseases or other conditions affecting the absorption, distribution, metabolism, and excretion of oral drugs.
8. Disagree to strict contraception within one year after the trial
9. Has any other conditions judged by the investigator as not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Recovery of total radioactivity in urine and fecal samples | up to 504 hours post dose
  Mass balance recovery of total radioactivity in urine and fecal samples
Total radioactivity in plasma PK: Cmax | up to 504 hours post dose
  Highest radioactivity observed plasma concentration
Total radioactivity in plasma PK: Area under the curve | up to 504 hours post dose
  Area under the plasma concentration time curve
Total radioactivity in plasma PK: t1/2 | up to 504 hours post dose
  Elimination half-life
Total radioactivity in plasma PK: MRT | up to 504 hours post dose
  Mean residence time
Total radioactivity in plasma PK: Tmax | up to 504 hours post dose
  Time for Cmax
Percentage of radioactivity and identification of metabolites in plasma, urine and fecal samples | up to 504 hours post dose
  Percentage of prototype drugs and its metabolites in plasma, urine and fecal samples. Identification of the major metabolites
Whole blood to plasma total radioactivity ratio | up to 504 hours post dose

SECONDARY OUTCOMES:
JAB-21822 PK: Cmax | up to 504 hours post dose
  Highest observed plasma concentration of JAB-21822
JAB-21822 PK: Area under the curve | up to 504 hours post dose
  Area under the plasma concentration time curve of JAB-21822
JAB-21822 PK: t1/2 | up to 504 hours post dose
  Elimination half-life of JAB-21822
JAB-21822 PK: MRT | up to 504 hours post dose
  Mean residence time of JAB-21822
JAB-21822 PK: Tmax | up to 504 hours post dose
  Time for Cmax of JAB-21822
Number of participants with adverse events | up to 504 hours post dose
  All subjects will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms and ophthalmological assessments

CONTACTS AND LOCATIONS:
Overall Officials: Miao Liyan doctor of pharmacy, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No